CLINICAL TRIAL: NCT04363346
Title: Study of FT516 Safety and Feasibility for the Treatment of Coronavirus Disease 2019 (COVID-19) in Hospitalized Patients With Hypoxia
Brief Title: Study of FT516 for the Treatment of COVID-19 in Hospitalized Patients With Hypoxia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IDIM-2020-28708; 2020LS083 (Other: University of Minnesota Masonic Cancer Center)
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
Keywords: COVID-19; Corona Virus; SARS-COV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: The study starts with a fast-track design by proceeding in cohorts of one patient until the first DLT is observed. If no DLT is observed, escalation continues by one patient per cohort until Dose Strategy 3 is reached. If the MTD is not yet established by Dose Strategy 3, Dose Strategy 3 is expanded to 6 patients using the final stage of a "3+3" design. An extension of 4 additional patients is planned if FT516 continues to be safe for a total of 10 patients treated at the MTD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Strategy 1 (Experimental): Dose Strategy 1:
  Day 1 - FT516 is given at 9x107 cells/dose (low)
  Interventions: Drug: FT516
- Dose Strategy 2 (Experimental): Dose Strategy 2:
  Day 1 - FT516 is given at 9x107 cells/dose (low) + Day 4 - FT516 is given at 3x108 cells/dose (mid)
  Interventions: Drug: FT516
- Dose Strategy 3 (Experimental): Dose Strategy 3:
  Day 1 - FT516 is given at 9x107 cells/dose (low) + Day 4 - FT516 is given at 3x108 cells/dose (mid) + Day 7 - FT516 is given at 9x108 cells/dose (high)
  Interventions: Drug: FT516

INTERVENTIONS:
Drug: FT516 — FT516 is an off-the-shelf cryopreserved NK cell product derived from an iPSC that was transduced with a high affinity, ADAM17 non-cleavable CD16 (Fc receptor) that maintains CD16 on the cell surface, which remains fully functional after NK cell activation.

SUMMARY:
This is a Phase I study with the primary objective of identifying the maximum tolerated dose (MTD) of FT516 using 3 dose-escalation strategies (number of doses and cell dose) for the treatment of coronavirus disease 2019 (COVID-19). This study provides initial estimates of safety and efficacy based on stable respiratory function, as well as, determining the feasibility for full-scale studies designed both for efficacy and safety.

DETAILED DESCRIPTION:
Given the urgency of COVID-19 and the known anti-viral activity of natural killer (NK) cells, this clinical trial uses immediately available off-the-shelf induced pluripotent stem cell (iPSC) derived NK cells already being used to treat cancer patients.

FT516 is an off-the-shelf cryopreserved NK cell product derived from an iPSC that was transduced with a high affinity, ADAM17 non-cleavable CD16 (Fc receptor) that maintains CD16 on the cell surface, which remains fully functional after NK cell activation. The investigators expect that natural developing anti-COVID IgG (early data suggest that some develop in 7-10 days after diagnosis) will enhance targeting of FT516 to infected cells.

ELIGIBILITY:
Inclusion Criteria:

* Has laboratory-confirmed novel coronavirus (SARS-CoV-2) infection as determined by polymerase chain reaction (PCR), or other commercial or public health assay.
* Requires hospitalization and meets the following:

  * Radiographic infiltrates by imaging (chest x-ray, CT scan)
  * Able to maintain Sp02 ≥ 93% oxygen supplementation to a maximum 4L by low flow O2-delivery device at rest
  * IL-6 level ≥40 pg/ml but <150 pg/mL OR CRP ≥40 mg/L (4 mg/dL) but <150 mg/L (15 mg/dL)
  * Ferritin < 1000 ng/mL
  * HCT-CI score of 4 or less - For this score, if PFTs results are not available, any patient requiring oxygen prior to COVID-19 illness is not eligible
* Report of usual daily activity level (before COVID-19 illness) of Karnofsky ≥70%
* ≥ 18 years of age, but < 76 years at time of consent signing
* Females of child-bearing potential and males with partners of child-bearing potential must agree to use highly effective contraception from the time of consent and for at least 3 months after the last dose of FT516
* Agrees to and signs the separate consent for up to 15 years of follow-up on a separate LTFU companion study (IDIM-2020-28770)
* Voluntary written consent prior to the performance of any research related procedures

Exclusion Criteria:

* Any medical condition or clinical laboratory abnormality that per Investigator judgement precludes safe participation in and completion of the study, or which could affect compliance with protocol conduct or interpretation of results.
* Need for higher-percentage oxygen delivery device (face mask, oxymizer, nonrebreather, venti-mask or pressure support with CPAP/BiPAP)
* Patients with adequate oxygenation on room air
* Receiving concomitant COVID-19 directed therapy (drugs may be stopped to make patients eligible)
* Known allergy to the following FT516 components: albumin (human) or DMSO
* Any known condition that requires systemic immunosuppressive therapy (> 5mg prednisone daily or equivalent) topical and inhale steroids are permitted
* Active autoimmune disease requiring systemic immunosuppressive therapy
* History of severe asthma and currently on chronic systemic medications (mild asthma requiring inhaled steroids only is eligible)
* Known history of HIV positivity
* Pregnant or breast feeding

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Number of participants with Dose Limiting Toxicity Events | within 7 days after the last dose of FT516
  An accelerated (fast-track) design will continue until first DLT is observed or the maximum Tolerated Dose (MTD) is determined.
  DLT is defined as any treatment emergent toxicity within 7 days after the last dose of FT516 meeting one of the following criteria based on CTCAE v5:
  * Grade 3 or greater infusion related reaction following FT516 infusion
  * Any new or worsening Grade 3 and any Grade 4 adverse events with the exception of the following known complications of COVID-19:
    * Grade 3 gastrointestinal disorders (diarrhea)
    * Grade 3 hepatic investigations (ALT increased, AST increased)
    * Grade 3 leukopenia/lymphopenia
  * Respiratory deterioration between the 1st dose and 7 days after the last dose of FT516 defined as the need for any type of assisted ventilation (invasive or non-invasive including BiPAP) or oxygen delivery device intended to deliver ≥60% FiO2 (including non-rebreather mask or >10L by simple facemask) to maintain an SpO2 >88%.

SECONDARY OUTCOMES:
The time in days from the 1st FT516 infusion to the elimination of viral shedding in nasal pharyngeal and stool samples | 36 days
The time in days from the 1st FT516 infusion to discontinued need for supplemental oxygen | 36 Days
The time in days from the 1st FT516 infusion to hospital discharge | 36 Days

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Joshua Rhein, MD, Principal Investigator — Department of Medicine, University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States